CLINICAL TRIAL: NCT01941277
Title: Effect of Exercise on Insulin Resistance
Acronym: EFFORT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: funding withdrawn
Sponsor: Alere San Diego (Industry)
Responsible Party: Sponsor
Organization: Abbott RDx Cardiometabolic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BSTE-0902
Record Dates: First submitted 2013-09-06; First posted 2013-09-13 (Estimated); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Prediabetic State
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive Exercise Group (Experimental): Behavioral
  Interventions: Behavioral: Intensive Exercise Group
- Current Recommendations Exercise Group (Experimental): Behavioral
  Interventions: Behavioral: Current Recommendations Exercise Group

INTERVENTIONS:
Behavioral: Current Recommendations Exercise Group
  Arms: Current Recommendations Exercise Group
Behavioral: Intensive Exercise Group
  Arms: Intensive Exercise Group

SUMMARY:
The purpose of this study is to evaluate the effect of exercise on Insulin Resistance (IR) in subjects who do not routinely exercise and who are at risk of developing diabetes (prediabetes).

It is estimated that approximately 30-90 people will participate in this study at three study sites in the United States and United Kingdom.

ELIGIBILITY:
Inclusion Criteria

1. Aged 18 to 75 years.
2. Meets one of the three diagnostic criteria listed below (based on screening results or recorded result within one week of enrollment);

   1. Fasting plasma or whole blood glucose (fasting defined as no caloric intake for at least 8 hours): 100 ≤ 125 mg/dL (6.0-6.9 mmol/L)
   2. HbA1c of 5.7% - 6.4% (39 - 46 mmol/mol)
   3. 2-hour plasma glucose of 140-199 mg/dL (7.8-11.0 mmol/L) during an OGTT (as described by the WHO using a glucose load of 75 g anhydrous glucose dissolved in water)
3. No clinically significant adverse exercise response during the maximal graded exercise test

Exclusion Criteria

1. Weight loss diet program or weight change (>10%) within the past 6 months
2. Daily physical activity of >10,000 steps per day (as measured during the interval between visits 1 and 2)
3. Participates in deliberate structured exercise
4. Pregnant or intending to become pregnant
5. Cognitive or intellectual disability that prevents subject from providing informed consent or following protocol instructions.
6. Unwillingness to participate in all study procedures
7. Inability to give blood through multiple venous phlebotomies or to have an intravenous catheter
8. BMI greater than 40 kg/m2
9. Concurrent participation in another lifestyle modification trial
10. Diagnosis of diabetes based on any one of the following criteria:

    1. Fasting plasma or whole blood glucose ≥ 126 mg/dL (7 mmol/L)
    2. HbA1c of >6.5% (>47 mmol/mol)
    3. 2-hour plasma glucose ≥ 200 mg/dL (11.1 mmol/L) during an OGTT
11. Any pre-existing or newly discovered medical condition that is deemed likely to put the subject at risk of injury during this trial. This may include but is not limited to:

    1. Clinically relevant vascular or cerebrovascular event (e.g. stroke, recurrent transient ischemic attack (TIA), deep venous thrombosis or intracardiac thrombi, clinically significant edema within the previous 6 months
    2. Current use of anti-psychotic, anti-convulsant, anti-coagulant, sedative medication, or cognition-enhancing medications
    3. Current use of beta blockers (beta-adrenergic blocking agents)
    4. Current or previous use (within the past year) of the following medications: diabetes related medications or insulin; metformin; growth hormone; glucagon; dipeptidyl peptidase-4(DPP-4) inhibitors (saxagliptin, stigagliptin); glucagon-Like Peptide-1(GLP-1) mimetics (exenatide, liraglutide); sulfonylurea medication or other potential confounding medications
    5. Medical conditon which predetermines insulin resistance (e.g. Marfan syndrome / severe Polycystic ovary syndrome (PCOS) / Cushing syndrome etc.).
    6. Fasting triglycerides > 1000 mg/dL.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
A decrease in Insulin Resistance (IR) as measured by a change in IR. | change between baseline and 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rick San George, PhD, Study Director — Alere San Diego; Michael Trenell, PhD, Principal Investigator — Newcastle University
Locations (2):
- United Kingdom (2):
  - Manchester University, Manchester
  - Move Lab, Newcastle upon Tyne